CLINICAL TRIAL: NCT04391114
Title: The Operative Parameters and Postoperative Outcomes of the Top-Down Holmium Laser Enucleation of the Prostate (HoLEP) Technique vs the Traditional HoLEP for Treatment of Benign Prostatic Hyperplasia (BPH): A Randomized Prospective Comparative Study
Brief Title: Top-Down Holmium Laser Enucleation of the Prostate (HoLEP) vs the Traditional HoLEP for Treatment of Benign Prostatic Hyperplasia (BPH)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thunder Bay Regional Health Research Institute (Other)
Responsible Party: Principal Investigator, Hazem Elmansy, Urology Surgeon, Thunder Bay Regional Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2019518
Record Dates: First submitted 2020-05-06; First posted 2020-05-18 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-08

CONDITIONS: Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Intervention Model Description: Prospective comparative randomized controlled trial comparing two standard of care treatments
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional HoLEP (Active Comparator): Holmium laser enucleation of the prostate (HoLEP), first reported by Fraundorfer et al in 1998, is a more recent step in the evolution of holmium laser prostatectomy. HoLEP is a safe and effective procedure which has demonstrated comparable results to Transurethral Resection of the Prostate (TURP) and open prostatectomy for patients with symptomatic enlarged prostate, with low morbidity and short hospital stay [4]. The improvement in outcome parameters is durable, and the late complications and reoperation rates reported are very low [5]. HoLEP is equally suitable for small, medium and larger prostate glands, with clinical outcomes that are independent of prostate size, unlike TURP. HOLEP offers patients the alterative of being treated endoscopically with minimal blood loss, short catheterization time, and decreased hospital stay [6].
  Interventions: Procedure: Traditional HoLEP
- Top-Down HoLEP (Active Comparator): The "Top-Down" HoLEP technique is a novel technique which offers potential benefits to the Traditional HoLEP procedure, including decreased complexity, a reduced learning curve, with anticipated improved continence [8]. A variation of this method is also being explored in Japan (termed the "en-bloc technique with anteroposterior dissection HoLEP") [9]. The main difference between the Top-Down and Traditional approach is that the direction of lateral dissection begins from upwards to downwards. This could help in avoiding the overtraction of the mucosal strip overlying the posterior urethral sphincter, which theoretically leads to a decrease in the incidence of postoperative stress incontinence. Moreover, using the Top-Down approach should lead to a decrease in the incidence of lost enucleation planes, which results in decreasing the intraoperative time and decreasing the number of cases required to master the HoLEP technique.
  Interventions: Procedure: Top-Down HoLEP

INTERVENTIONS:
Procedure: Traditional HoLEP — Holmium laser enucleation of the prostate (HoLEP), first reported by Fraundorfer et al in 1998, is a more recent step in the evolution of holmium laser prostatectomy. HoLEP is a safe and effective procedure which has demonstrated comparable results to TURP and open prostatectomy for patients with symptomatic enlarged prostate, with low morbidity and short hospital stay [4]. The improvement in outcome parameters is durable, and the late complications and reoperation rates reported are very low [5]. HoLEP is equally suitable for small, medium and larger prostate glands, with clinical outcomes that are independent of prostate size, unlike TURP. HOLEP offers patients the alterative of being treated endoscopically with minimal blood loss, short catheterization time, and decreased hospital stay [6].
  Arms: Traditional HoLEP
Procedure: Top-Down HoLEP — The main difference between the Top-Down and Traditional approach is that the direction of lateral dissection begins from upwards to downwards. This could help in avoiding the overtraction of the mucosal strip overlying the posterior urethral sphincter, which theoretically leads to a decrease in the incidence of postoperative stress incontinence. Moreover, using the Top-Down approach should lead to a decrease in the incidence of lost enucleation planes, which results in decreasing the intraoperative time and decreasing the number of cases required to master the HoLEP technique.
  Arms: Top-Down HoLEP

SUMMARY:
Benign prostatic hyperplasia (BPH), the non-malignant enlargement of the prostate gland, places pressure on the urethra and causes urination difficulties and bladder problems. Lower Urinary Tract Symptoms (LUTS) secondary to BPH is a common condition in aging men, with an overall prevalence of more than 50% in those older than 50 years of age. Men with LUTS often experience sexual dysfunction including ejaculatory loss, painful ejaculation, and erectile dysfunction, which among other complications can also lead to a decreased quality of life.

Holmium laser enucleation of the prostate (HoLEP), first reported by Fraundorfer et al in 1998, is a more recent step in the evolution of holmium laser prostatectomy. HOLEP offers patients the alternative of being treated endoscopically with minimal blood loss, short catheterization time, and decreased hospital stay.

One noted drawback to HoLEP, and the primary reason why it has yet to become the new standard for treatment of symptomatic BPH, is the complexity of this procedure, with a prolonged learning curve. Modifications to the procedure have thus been explored in order to address this limitation. The "Top-Down" HoLEP technique is a novel technique which offers potential benefits to the Traditional HoLEP procedure, including decreased complexity, a reduced learning curve, with anticipated improved continence.

This study will compare the operating time between the Top-Down Holmium Laser Enucleation of the prostate (HoLEP) and the Traditional HoLEP for the treatment of patients with symptomatic bladder outlet obstruction due to BPH in Northwestern Ontario.

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH), the non-malignant enlargement of the prostate gland, places pressure on the urethra and causes urination difficulties and bladder problems. Lower Urinary Tract Symptoms (LUTS) secondary to BPH is a common condition in aging men, with an overall prevalence of more than 50% in those older than 50 years of age. Men with LUTS often experience sexual dysfunction including ejaculatory loss, painful ejaculation, and erectile dysfunction, which among other complications can also lead to a decreased quality of life.

Conventional Transurethral Resection of the Prostate (TURP), a surgical technique in which excess prostate tissue is removed using a resectoscope, remains the gold standard treatment in most centres for symptomatic BPH. However, morbidity after TURP is high, especially bleeding requiring blood transfusion (0.4-6.4%) and late postoperative bleeding (1.3-1.7%).

Holmium laser enucleation of the prostate (HoLEP), first reported by Fraundorfer et al in 1998, is a more recent step in the evolution of holmium laser prostatectomy. HoLEP is a safe and effective procedure which has demonstrated comparable results to TURP and open prostatectomy for patients with symptomatic enlarged prostate, with low morbidity and short hospital stay. The improvement in outcome parameters is durable, and the late complications and reoperation rates reported are very low. HoLEP is equally suitable for small, medium and larger prostate glands, with clinical outcomes that are independent of prostate size, unlike TURP. HOLEP offers patients the alternative of being treated endoscopically with minimal blood loss, short catheterization time, and decreased hospital stay.

One noted drawback to HoLEP, and the primary reason why it has yet to become the new standard for treatment of symptomatic BPH, is the complexity of this procedure, with a prolonged learning curve as compared to TURP. Modifications to the procedure have thus been explored in order to address this limitation. The "Top-Down" HoLEP technique is a novel technique which offers potential benefits to the Traditional HoLEP procedure, including decreased complexity, a reduced learning curve, with anticipated improved continence. A variation of this method is also being explored in Japan (termed the "en-bloc technique with anteroposterior dissection HoLEP"). The main difference between the Top-Down and Traditional approach is that the direction of lateral dissection begins from upwards to downwards. This could help in avoiding the overtraction of the mucosal strip overlying the posterior urethral sphincter, which theoretically leads to a decrease in the incidence of postoperative stress incontinence. Moreover, using the Top-Down approach should lead to a decrease in the incidence of lost enucleation planes, which results in decreasing the intraoperative time and decreasing the number of cases required to master the HoLEP technique.

In a recent retrospective review of this technique in Indiana, promising early operative results in a small sample size were demonstrated. The mean enucleation time and mean enucleation rate were both faster when comparing the 49 patients who underwent the top-down technique as compared to those 37 patients who underwent the traditional HoLEP technique. While the results of this particular study are limited by the relatively small number of cases and retrospective nature of the study, the potential value of this technique is evident. A retrospective review of 26 patients who underwent surgery using the en-bloc technique in Japan led to similar conclusions regarding the complexity of the procedure and improvement of rates. While this procedure demonstrates potential over the conventional TURP treatment and traditional HoLEP treatment of symptomatic BPH, the specific techniques of the Top-down technique must be further explored.

Our most recent online publication about Top-Down HoLEP early outcomes in 60 patients who underwent HoLEP between 2017 and 2018 with median prostate volume of 124ml (70-266) demonstrated at 3 months follow-up, the urine stream significantly improved with a median Qmax 23.6 mL/s (17-42). Two patients (3.3%) had urge incontinence, and 2 other patients (3.3%) had stress incontinence at 3 months follow-up.

This study will compare the operating time between the Top-Down Holmium Laser Enucleation of the prostate (HoLEP) and the Traditional HoLEP for the treatment of patients with symptomatic bladder outlet obstruction due to BPH in Northwestern Ontario.

ELIGIBILITY:
Inclusion Criteria:

1. Males over 50 years of age at the time of enrollment
2. Referred to urology for refractory LUTS secondary to BPH
3. Failed medical (non-surgical) treatment
4. Prostate size on preoperative TRUS of > 80 ml
5. IPSS >15, QOL score ≥3 and Qmax <15 ml/sec
6. Written informed consent to participate in the study
7. Ability to comply with the requirements of the study procedures

Exclusion Criteria:

1. Previous surgical treatment for BPH
2. Presence of bladder stones
3. History of prostate cancer
4. Prostate size < 80 mL
5. History of urethral stenosis or its management
6. Known or suspected neurogenic bladder
7. Participants with active urinary tract infection until appropriately treated
8. Participants with preexisting conditions, which, in the opinion of the investigator, interfere with the conduct of the study
9. Participants who lack the capacity, or cannot speak English, in order to provide free and informed written consent

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Operating time | Operating time/Surgery
  Length of time required for surgical procedure

SECONDARY OUTCOMES:
Intraoperative adverse events | During surgery
  Incidence of bleeding and blood transfusion; and operative time/laser time ratio to be investigated
Length of hospital stay | 1-day post-op
  Time participant had to remain in hospital following surgery. Time to be measured in hours and minutes
Time to catheter removal | 1-day post-op
  Time until catheter was removed from participant post-surgery. Measured in hours and minutes
International Prostate Symptom Scores (I-PSS) | 1-year post-op
  The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic).
Quality of Life (QoL) scores | 1-year post-op
  One question asking; "If you were to spend the rest of your life with your urinary condition just the way it is now, how would you feel about that? Scored from 0-6 with 0 being "delighted" and 6 being "terrible". Higher the score, the lower the quality of life.
peak urine flow rates (Qmax) | 1-year post-op
  Indicates the maximum urine flow rate. In men peak flow rates (Qmax) greater than 15-20 ml/second are considered normal, rates less than 10 ml/second are considered abnormal. This is measured by Uroflowmetry, also called a uroflow test, which measures the flow and force of urine stream during urination.
post-void residual urine volume (PVR) | 1-year post-op
  The amount of urine retained in the bladder after a voluntary void. Incomplete bladder emptying is diagnosed by postvoid catheterization or ultrasonography showing an elevated residual urine volume. A volume < 50 mL is normal; <100 mL is usually acceptable in patients > 65 but abnormal in younger patients

CONTACTS AND LOCATIONS:
Overall Officials: Hazem Elmansy, MD, Principal Investigator — Thunder Bay Regional Health Sciences Centre
Locations (1):
- Thunder Bay Regional Health Sciences Centre/Thunder Bay Regional Health Research Institute, Thunder Bay, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We have no plan to share individual data with any other researchers. We do plan to present our findings at various national and international conferences in the future... however all participant data will have been de-identified and grouped at that point.